CLINICAL TRIAL: NCT04361357
Title: The Effects of Enteral Whey Protein Supplement on Serum Albumin Level in Acute Critically Ill Neurological Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: zhangyan
Record Dates: First submitted 2020-03-05; First posted 2020-04-24 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-02

CONDITIONS: Nutrition Disorders; Neurologic Disorder
Keywords: critically ill neurological disease; whey protein; nutrition; acute phase
MeSH Terms: conditions — Nutrition Disorders; Nervous System Diseases | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): whey protein powder was added on the basis of standardized enteral nutrition preparation.
  Interventions: Other: whey protein
- Control group (No Intervention): standardized enteral nutrition preparation only.

INTERVENTIONS:
Other: whey protein — whey protein powder was added on the basis of standardized enteral nutrition preparation.
  Arms: Experimental group

SUMMARY:
The incidence of malnutrition in patients with severe neurological diseases is approximately 37%, among which hypoproteinemia is a common manifestation. It has been confirmed that serum albumin level is closely related to severity and mortality for patients. Protein is the basic component of tissue cells in the body, which plays an important role in the growth and development of senescent cells and the repair of damaged tissues. At present, the results of some randomized controlled studies show that it is difficult to achieve enough protein supplementation by commercial standard enteral nutrition agents alone, and additional protein supplementation is required. Commercial standard enteral nutrition preparations, whose whole protein components are casein and soy protein, do not achieve optimal uptake and utilization compared to whey proteins, which are more readily absorbed and utilized by the human gut. Whey protein and its hydrolyzed products have better nutritional quality than casein, which can provide high-quality nitrogen source for enteral nutrition and play an important role in correcting negative nitrogen balance, promoting wound healing and improving body immunity. Whether whey protein supplementation based on standard enteral nutrition preparation can improve serum albumin level and reduce the incidence of hypoproteinemia in patients with severe acute neurological disease has not been proved. In conclusion, we propose the hypothesis that compared with the standard enteral nutrition preparation regimen, the enteral nutrition regimen supplemented with whey protein in patients with severe neurological disease is more beneficial to improve the nutritional indicators of patients and reduce the occurrence of hypoproteinemia. It is expected that this randomized controlled trial will provide a new clinical basis for optimizing the enteral nutrition support program for patients with severe neurological diseases.

DETAILED DESCRIPTION:
The purpose of the study is to compare standard enteral nutrition regimen with the enteral nutrition regimen supplemented with whey protein in severe neurological disease patients and to observe nutritional indicators improvement in these patients. A total of 116 subjects will be included. Counting process is as follows: referring available literature and the mean value of serum albumin in patients on the 14th day of our preliminary tests, and the difference test is used to compare the mean values of two independent samples. The ratio of the experimental group and control group is 1:1. It was assumed that the serum albumin level in the experimental group was higher than that in the control group. A single end is taken, α=0.05, 1-β=0.80, experimental group patients serum albumin（Χ±S）=37.9±5.1, the control group serum albumin（Χ±S）=35.6±4.8, so the total sample size was 116.It was estimated that 116 patients were enrolled consecutively, which were divided into experimental group and control group by computer generated random number table. Patients in both groups received enteral nutrition therapy with continuous tube feeding for 14 days. According to the nutritional treatment requirements of critically ill patients in the Asia-Pacific region in 2016, patients with severe acute stress were given energy demand for 25~30kcal/kg/d, protein demand for 1.2~2g/kg/d and other standardized clinical treatments. Control group nutrition program: standardized enteral nutrition preparation only. Experimental group nutrition program: whey protein powder was added on the basis of standardized enteral nutrition preparation. According to the body weight of the patients, different enteral nutritional preparations and dose adjustments were selected to ensure that the calorie and protein intake of the two groups of patients met the above nutritional treatment requirements.Primary endpoint: serum albumin level at 14 days of enteral nutrition. Secondary end points: 1. APACHE II, GCS and other clinical scores at 14 days; 2. total serum protein, proalbumin, hemoglobin and other nutritional indicators; 3. the number and ratio of white blood cells, neutrophils, c-reactive protein, interleukin-6, procalcitonin, absolute count of T lymphocyte subsets, immunoglobulin and other inflammatory indicators at 14 days; 4. the number of cases of gastrointestinal complications such as gastric retention, vomiting, diarrhea, abdominal distention, constipation and gastrointestinal bleeding during the 14 days of enteral nutrition; 5. the number of patients with serum albumin < 30g/L within 14 days after admission.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of severe neurological Disease
2. Serum albumin ≥30g/L
3. Weight: 50~90kg
4. Nutrition risk screening 2002 (NRS2002) ≥3 points
5. Acute gastrointestinal function injury (acute gastrointestinal injury, AGI) class 1~2
6. Expected enteral nutrition in tube feeding for at least 14 days
7. Obtain the informed consent of the patient or its authorized client

Exclusion Criteria:

1. Pregnant and breast-feeding women
2. Serious heart, lung and other important organ function injury
3. Malignant tumor
4. Hypothermia treatment
5. BMI≥28
6. Allergic to milk
7. Receiving parenteral nutritional support therapy
8. APACHE II ≥30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum albumin level | At 14 days of enteral nutrition

SECONDARY OUTCOMES:
Serum proalbumin level | At 14 days of enteral nutrition

OTHER OUTCOMES:
The number of gastrointestinal complications | During the 14 days of enteral nutrition
  such as gastric retention, vomiting, diarrhea, abdominal distention, constipation and gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Su, MD, Study Director — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
study protocol can be shared.
Supporting Information: Study Protocol
Time Frame: after Dec 2020, always
Access Criteria: email to authors